CLINICAL TRIAL: NCT05965128
Title: Promotion and Application of a New Three-level Etiological Diagnosis Strategy for Fever Clinics in Respiratory Infectious Diseases
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: KY2022-955
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Infectious Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Relying on fever clinics, this project evaluates the clinical diagnostic efficiency of the three-level pathogen diagnostic system, monitors changes in respiratory pathogens, and realizes real-time monitoring and early warning of acute respiratory infectious diseases in Shanghai.

DETAILED DESCRIPTION:
This study mainly includes subjects who enter the outpatient and emergency departments, fever clinics, and wards of each center from December 2022. According to the clinical manifestations and epidemiological information of the patients, different step-by-step detection methods will be adopted to optimize the allocation of clinical resources and improve the quality of life. This study aims to improve pathogen diagnosis efficiency and achieve regional respiratory early warning.

ELIGIBILITY:
Inclusion Criteria:

1. Acute onset within one week;
2. 18-70 years old;
3. Present with pneumonia (present with pulmonary signs or radiological changes) or influenza-like illness (including the following symptoms: sudden onset of fever (>38 ℃),plus cough and/or other respiratory symptoms such as shortness of breath plus one or more systemic symptoms (fatigue, headache ect.))

Exclusion Criteria:

1. Unable to collect nasal/nasopharyngeal swab/wash/aspirate due to structural disorder or mental problem.
2. Patients with psycological problem or unconsciousness who cannot tell the disease history and cooperate with medical examinations;

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: this study enrolled patients who were admitted to the fever clinics and emergency room for influenza-like illness or pneumonia and pathogenic detection was necessary for clincial diagnosis and treatment.
Sampling Method: Probability Sample
Enrollment: 1255 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the detectioin rate of pathogenic microorganism in each step | 48 hours
  the detectioin rate of pathogenic microorganism in each step

SECONDARY OUTCOMES:
hospitalization rate | 48 hours
  hospitalization rate
rate of critical illness | 48 hours
  rate of critical illness

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Heilongjiang Provincial Hospital, Harbin, Heilongjinag
  - People's Hospital of Inner Mongolia Autonomous Region, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shenyang Sixth People's Hospital, Shenyang, Liaoning
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Jining Public Health Center, Jining, Shandong
  - Fudan University Affiliated Huashan Hospital, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Ruian City People's Hospital, Rui’an, Zhejiang

IPD SHARING:
Plan to Share IPD: No